CLINICAL TRIAL: NCT06621758
Title: Communication Regarding Preclinical Dementia Diagnostic and Diagnostic Disclosure Among Patients with MCI and SCD
Status: Not yet recruiting | Type: Observational
Sponsor: Danish Dementia Research Centre (Network)
Collaborators: Toulouse University Hospital, Department of Geriatric & Internal Medicine, France (Unknown); Universitair Ziekenhuis Brussel, Department of Neurology, Belgium (Unknown); University Medical Centre Ljubljana, Department of Neurology, Slovenia (Unknown)
Responsible Party: Principal Investigator, Kristian Steen Frederiksen, MD, MD, PhD, clinical lector, Danish Dementia Research Centre
Other Study IDs: F-24061891; ERA PerMed JTC2021 (Other: European Commission)
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment (MCI); Subjective Cognitive Decline (SCD)
Keywords: communication; biomarkers; counseling; diagnostic disclosure; MCI; SCD
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Communication | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MCI: Individuals diagnosed with mild cognitive impairment (MCI)
  Interventions: Other: questionnaire
- SCD: Individuals diagnosed with subjective cognitive decline (SCD)
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — Questionnaire regarding biomarker counseling and diagnostic disclosure

SUMMARY:
The study investigate what information individuals with SCD or MCI and their co-participant would like to receive during pre-diagnostic counseling and diagnostic disclosure, and how this information should be conveyed.

DETAILED DESCRIPTION:
Improved diagnostic work-up and the introduction of disease-modifying treatment have led to a shift towards earlier diagnosis. However, there are a need for better understanding of how best to communicate about biomarker use, assessment, and results in individuals with subjective cognitive decline (SCD) and mild cognitive impairment (MCI).

Objective:

The overarching objective of this study is:

To understand what information individuals with SCD or MCI and their co-participant would like to receive during pre-diagnostic counseling and diagnostic disclosure, and how this information should be conveyed.

Methods: a prospective survey study Persons diagnosed with SCD or MCI and co-participants will be recruited consecutively from the memory clinic, Copenhagen University Hospital - Rigshospitalet (Denmark), Toulouse University Hospital, (France), University Medical Centre Ljubljana (Slovenia) and Universitair Ziekenhuis Brussel (Belgium)

Approximately 30 persons and respective co-participants will be included from each hospital over a period of 12 months.

Each participating person and co-participant will be asked to complete a very brief questionnaire immediately after disclosure of the diagnosis, and another questionnaire 2-6 weeks after the disclosure visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with SCD or MCI
* Lumbar puncture performed during the diagnostic process
* Age at or below 80 years
* MMSE at or above 24

Exclusion Criteria:

* Diagnosis of current major psychiatric disorder (schizophrenia, bipolar disorder, psychosis)
* Current excessive alcohol intake or substance abuse

Inclusion criteria for the co-participant:

* Attended the diagnostic disclosure visit together with the individual diagnosed with SCD or MCI

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with SCD or MCI and co-participants will be recruited consecutively from the memory clinic, Copenhagen University Hospital - Rigshospitalet (Denmark), Toulouse University Hospital, (France), University Medical Centre Ljubljana (Slovenia) and Universitair Ziekenhuis Brussel (Belgium)
  Approximately 30 persons and respective co-participants will be included from each hospital.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Important issues in communication | From enrollment to the second questionnaire after 6 weeks
  Rating of which issues are important for persons with SCD or MCI and their co-participant in the pre-diagnostic counseling and diagnostic disclosure communication.

IPD SHARING:
Plan to Share IPD: Undecided